CLINICAL TRIAL: NCT01118689
Title: A Phase I, Open Label, Dose Escalation Study of Oral Administration of Single Agent MLN0128 in Subjects With Relapsed or Refractory Multiple Myeloma or Waldenstrom Macroglobulinemia
Brief Title: Dose Escalation Study of MLN0128 in Relapsed or Refractory Multiple Myeloma or Waldenstrom Macroglobulinemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INK-128-002
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN0128 (Experimental)
  Interventions: Drug: MLN0128

INTERVENTIONS:
Drug: MLN0128 — MLN0128 administered orally once daily for 28 days

SUMMARY:
The purpose of this study is to determine the safety, tolerability, maximum tolerated dose and pharmacokinetics of MLN0128 in patients with Relapsed or Refractory Multiple Myeloma or Waldenstrom Macroglobulinemia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, including males and females;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2;
* Life expectancy of ≥3 months;
* Does not have diabetes and has normal fasting serum glucose and fasting triglycerides ≤ 300 mg/dL
* For women of child-bearing potential, negative serum pregnancy test within 14 days prior to the first study drug administration and use of physician-approved method of birth control from 30 days prior to the first study drug administration to 30 days following the last study drug administration;
* Male subjects must be surgically sterile or must agree to use physician-approved contraception during the study and for 30 days following the last study drug administration;
* Ability to swallow oral medications;
* Ability to understand and willingness to sign informed consent form prior to initiation of any study procedures;

Exclusion Criteria:

* Have received prior cancer therapy or other investigational therapy within 2 weeks prior to the first administration of study drug.
* Known impaired cardiac function or clinically significant cardiac disease
* HIV infection;
* Failed to recover from the reversible effects of prior anticancer therapies:
* Pregnancy (positive serum or urine pregnancy test) or breast feeding;
* Malabsorption due to prior gastrointestinal (GI) surgery, GI disease;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
determine the dose limiting toxicities | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - San Francisco, California
  - Denver, Colorado
  - Boston, Massachusetts
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Nashville, Tennessee